CLINICAL TRIAL: NCT03896022
Title: Auriculotherapy as an Adjunct for Pain Management During First Trimester Vacuum Aspiration Abortion: a Randomized, Double-blinded, Three Arm Trial
Brief Title: Auriculotherapy - Pain Management of Aspiration Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Carolyn Westhoff, Professor of Obstetrics and Gynecology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AAAS0917
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Results first posted 2021-01-22 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Abortion in First Trimester
Keywords: auriculotherapy; abortion; pain management
MeSH Terms: conditions — Agnosia | interventions — Acupressure; Acupuncture Therapy; Needles

STUDY DESIGN:
Intervention Model Description: This 3-arm randomized trial will assign participants 1:1:1 to receive either of two active treatments (acupressure or acupuncture) or placebo (inert adhesive disks applied to ears).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A designated investigator (auriculotherapy provider) will apply the intervention prior to the aspiration abortion; thus the care provider (abortion provider) will not be aware of the treatment arm.
  Participant will wear a surgical hat that covers their ears and the adhesive disks appear similar for the treatments and the placebo arm; thus the participants will be unaware of their treatment assignment.
  The research assistant collecting the outcomes data will not know which treatment arm the participant belongs to.
  Finally, treatment assignment will be coded in the study database until analysis is complete, so that the investigator will be unaware of the treatment assignment until analysis is complete and then un-blinding will occur.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Auriculotherapy - Acupressure with Gold Beads (Active Comparator): A designated trained auriculotherapy provider will place gold beads at five acupoints on each ear (10 points total). The beads are affixed with a small round adhesive disk. The beads will stay in place during the aspiration abortion and will be removed before the participant is discharged home.
  Interventions: Device: Acupressure with Beads
- Auriculotherapy - Acupuncture with Pyonex Needles (Active Comparator): A designated trained auriculotherapy provider will place 1.2mm (Pyonex) needles at five acupoints on each ear (10 points total). The needles are affixed with a small round adhesive disk. The needles will stay in place during the aspiration abortion and will be removed before the participant is discharged home.
  Interventions: Device: Acupuncture with Needles
- Placebo Group (Sham Comparator): A designated trained auriculotherapy provider will place adhesive disks at five acupoints on each ear (10 points total). The disks resemble those used with the active treatments. The disks will stay in place during the aspiration abortion and will be removed before the participant is discharged home.
  Interventions: Device: Placebo Adhesive Disks

INTERVENTIONS:
Device: Acupressure with Beads — Single-use gold-plated 1.2mm beads/balls attach to pre-specified acupoints on the participant's ears with adhesive disk/tape.
  Other Names: Accu-patch Pellets; Accu-patch Beads
  Arms: Auriculotherapy - Acupressure with Gold Beads
Device: Acupuncture with Needles — Single-use 1.2mm acupuncture press needles attach to pre-specified acupoints on the participant's ears with adhesive disk/tape.
  Other Names: Pyonex Needles; Seirin Pyonex Singles
  Arms: Auriculotherapy - Acupuncture with Pyonex Needles
Device: Placebo Adhesive Disks — Single-use adhesive disks without needles or beads.
  Other Names: Placebo Disks
  Arms: Placebo Group

SUMMARY:
Primary Objective: To assess whether usual care plus auricular acupressure with beads reduces subject-reported maximum pain during first trimester vacuum aspiration compared to usual care plus placebo.

Secondary Objective: To assess whether usual care plus auricular acupuncture with Pyonex™ needles reduces subject-reported maximum pain during first trimester vacuum aspiration as compared to usual care plus placebo. This assessment will replicate the previous trial and strengthen the evidence that auricular acupuncture is beneficial for aspiration abortion pain

Exploratory Objective: To assess whether usual care plus either auricular acupressure with beads or auricular acupuncture with Pyonex™ needles reduces subject-reported anxiety scores during first trimester vacuum aspiration as compared to women receiving usual care plus placebo.

DETAILED DESCRIPTION:
Most first trimester aspiration abortions are performed in the outpatient setting with a paracervical block and nonsteroidal anti-inflammatory drugs (NSAIDs) as the only analgesics. Yet first trimester aspiration pain control is often inadequate with 26-32% of women reporting that they experienced severe pain. Moderate sedation and general anesthesia are not readily available, and investigations on opioids and anxiolytics have consistently found them ineffective for first trimester aspiration abortion pain. In 2018, The National Academies of Sciences, Engineering, and Medicine (NASEM) recommended research to improve pain relief. Limited data indicate that acupuncture is valuable in dysmenorrhea and for labor pain, conditions in which pain may be similar to that experienced during aspiration abortion.

This randomized trial will recruit women seeking first trimester aspiration abortion. This study will evaluate two types of auriculotherapy applied to selected acupoints on the external ear. The study treatments are acupressure using gold beads and acupuncture using Pyonex needles; both are applied to the ear using adhesive disks. A control group will receive the adhesive disks alone. All participants will receive usual care for their aspiration abortion procedure, including a paracervical block and ibuprofen for pain management. The investigators will query the participants regarding pain and anxiety immediately after their procedure, in person, on the day of their procedure.

ELIGIBILITY:
bullets

Inclusion Criteria:

* Pregnant up to 13 weeks gestation
* Seeking aspiration abortion for any first trimester induced abortion, abnormal pregnancy, early pregnancy loss, retained products of conception, or molar pregnancy
* English- or Spanish-speaking
* Willingness to be randomized into one of the three arms.

Exclusion Criteria:

* Allergy to adhesives or gold
* Allergy or intolerance to ibuprofen or 1% lidocaine (paracervical block)
* Congenital anomaly or infection of the ear.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 177 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Westhoff, MD, MSc, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ndubisi C, Danvers A, Gold MA, Morrow L, Westhoff CL. Auricular acupuncture as an adjunct for pain management during first trimester abortion: a randomized, double-blinded, three arm trial. Contraception. 2019 Mar;99(3):143-147. doi: 10.1016/j.contraception.2018.11.016. Epub 2018 Dec 7. PMID 30529393

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 177 participants were randomized. 4 participants were excluded from the acupressure group (1 withdrew from the study after randomization and 3 did not have a procedure that day). The final analysis included 173 participants: 70 participants in the acupressure group, 51 in the acupuncture group, and 52 in the placebo group.
Period: Overall Study
Arm/Group | Auriculotherapy - Acupressure With Gold Beads | Auriculotherapy - Acupuncture With Pyonex Needles | Placebo Group
Started | 74 | 51 | 52
Completed | 70 | 51 | 52
Not Completed | 4 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Did not have procedure | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 177 participants were randomized. 4 participants were excluded from the acupressure group (1 withdrew from the study after randomization and 3 did not have a procedure that day). The final analysis included 173 participants: 70 participants in the acupressure group, 51 in the acupuncture group, and 52 in the placebo group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Auriculotherapy - Acupressure With Gold Beads | Auriculotherapy - Acupuncture With Pyonex Needles | Placebo Group | Total
Number analyzed (Participants) | 70 | 51 | 52 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (6.6) | 31.5 (6.2) | 30.3 (6.2) | 31.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 51 | 52 | 173
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 55 | 33 | 42 | 130
  Non-Hispanic White | 4 | 4 | 4 | 12
  Non-Hispanic Black | 8 | 9 | 2 | 19
  Other (Asian) | 3 | 5 | 2 | 10
  Unknown | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 51 | 52 | 173

OUTCOME MEASURES:

1. Primary Outcome: Pain Visual Analog Scale Score (Beads vs Placebo)
Description: Self-assessed maximum pain reported using a 0-100mm visual analog scale, where 100 signifies maximum pain. To measure pain experienced during aspiration abortion.
Time Frame: Immediately following the aspiration abortion procedure (approximately 10 minutes)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Auriculotherapy - Acupressure With Gold Beads | Placebo Group
Number analyzed (Participants) | 70 | 52
score on a scale | 50 [23 to 75.5] | 47.5 [31.3 to 73]

2. Secondary Outcome: Pain Visual Analog Scale Score (Needles vs Placebo)
Description: as for outcome 1
Time Frame: Immediately following the aspiration abortion procedure (approximately 10 minutes)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Auriculotherapy - Acupuncture With Pyonex Needles | Placebo Group
Number analyzed (Participants) | 51 | 52
score on a scale | 55 [28 to 78] | 47.5 [31.3 to 73]

3. Other Pre Specified Outcome: Anxiety Visual Analog Scale Score
Description: Self-assessed maximum anxiety reported using a 0-100 mm visual analog scale, where 100 signifies maximum anxiety. To measure anxiety during aspiration abortion.
Time Frame: Immediately following the aspiration abortion procedure (approximately 10 minutes)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Auriculotherapy - Acupressure With Gold Beads | Auriculotherapy - Acupuncture With Pyonex Needles | Placebo Group
Number analyzed (Participants) | 70 | 51 | 52
score on a scale | 26 [12.8 to 50] | 28 [10 to 65] | 21 [0 to 56]

ADVERSE EVENTS:
Time Frame: During and immediately following the aspiration abortion procedure (approximately 10 minutes).
Arm/Group | Auriculotherapy - Acupressure With Gold Beads | Auriculotherapy - Acupuncture With Pyonex Needles | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/51 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/51 | 0/52
Other Adverse Events (participants affected / at risk) | 0/70 | 0/51 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT03896022/Prot_SAP_000.pdf